CLINICAL TRIAL: NCT07046611
Title: Efficacy of Combined Ketamine and Levetiracetam as a Second-line Anti-seizure Medication for Generalized Convulsive Status Epilepticus in Children
Brief Title: Ketamine and Levetiracetam as Second-line Antiseizure Medication for Status Epilepticus in Children
Acronym: KLaSSEC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelkreem, Assistant Professor of Pediatrics, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Soh-Med-25-6-2PD
Record Dates: First submitted 2025-06-20; First posted 2025-07-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Generalized Convulsive Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Ketamine; Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine + Levetiracetam (Experimental)
  Interventions: Drug: Ketamine; Drug: Levetiracetam
- Placebo + Levetiracetam (Placebo Comparator)
  Interventions: Drug: Levetiracetam; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Intravenous ketamine (5 mg/ml concentration) 2 mg/kg (max 90 mg) over 2 minutes
  Arms: Ketamine + Levetiracetam
Drug: Levetiracetam — Intravenous levetiracetam (50 mg/ml concentration) 60 mg/kg (max 4500 mg) over 5 minutes
Drug: Placebo — Intravenous isotonic saline 0.4 mL/kg (maximum 18 mL) over 2 minutes
  Arms: Placebo + Levetiracetam

SUMMARY:
About 40% of children with generalized convulsive status epilepticus (GCSE) are not terminated by first-line benzodiazepines (BDZs), and approximately 50% of BDZ-refractory GCSE are not controlled by second-line antiseizure medications. This study investigates the efficacy of ketamine-levetiracetam combination vs. levetiracetam alone for treating children with BDZ-refractory GCSE.

DETAILED DESCRIPTION:
Generalized convulsive status epilepticus (GCSE) is the most common pediatric neurological emergency. Benzodiazepines (BDZs) are the recommended first-line anti-seizure medication (ASM) for GCSE, but they fail to halt seizures in about 40% of cases. Moreover, approximately 50% of BDZ-refractory GCSE are not terminated by second-line ASMs, including levetiracetam, valproate, and phenytoin. Continuous GCSE for a longer duration is associated with progressive brain injury and a higher risk of mortality, epilepsy, and permanent neurodevelopmental impairment. Therefore, early control of GCSE is pivotal for improving patients' outcomes.

A potential approach for early control of GCSE is the use of early ASM polytherapy. Ketamine is a promising option to be combined with standard ASMs for more rapid control of seizures. Ketamine has been used for decades for pediatric procedural analgosedation due to its excellent safety profile and wide therapeutic index. Ketamine works as a noncompetitive antagonist for N-methyl-D-aspartate (NMDA) receptors, which are progressively upregulated by way of receptor trafficking during ongoing seizure activity. Ketamine administration is associated with termination or attenuation of refractory SE (RSE) and super-refractory SE (SRSE). Multiple observational studies have reported the efficacy of ketamine in the pre-hospital emergency treatment of BZD-refractory status epilepticus. Furthermore, the recently published Ket-Mid study demonstrated that the ketamine-midazolam combination was more effective than midazolam alone in the initial treatment of pediatric GCSE. However, the value of combining ketamine with levetiracetam for the treatment of BZD-refractory status epilepticus has not been well investigated.

The present study (Ketamine and Levetiracetam as Second-line antiseizure medication for Status Epilepticus in Children, KLaSSEC) aims to investigate the efficacy of ketamine-levetiracetam combination vs. levetiracetam alone for treating children with BDZ-refractory GCSE. The findings could help earlier control of seizures and better clinical outcomes for children with status epilepticus

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 year to 16 years.
* Generalized convulsive status epilepticus (GCSE), defined as clinically observed generalized tonic-clonic convulsions that continue or recur without complete regaining of consciousness in between for longer than 5 minutes.
* Benzodiazepine-refractory, defined as continuous or recurrent GCSE in the emergency room after receiving an adequate benzodiazepine dose, with the last dose administered within 5 to 30 minutes.

Exclusion Criteria:

* Failure to obtain informed consent.
* Prior treatment with antiseizure medication or anticonvulsant sedatives other than benzodiazepines for the presenting GCSE episode.
* Endotracheal intubation before enrollment.
* Acute traumatic brain injury.
* Cardiac arrest/post-anoxic seizures
* Hypoglycemia or hyperglycemia.
* Known allergies or contraindications to ketamine or levetiracetam
* Failure to obtain intravenous access.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cessation of seizures at 20-minute | 20 minutes
  Number of participants with cessation of clinically evident seizures at 20-minute after starting study drug administration without endotracheal intubation or need for other antiseizure medications or anticonvulsant sedatives

SECONDARY OUTCOMES:
Number of participants with cessation of seizures at 5-minute | 5 minutes
  Number of participants with cessation of clinically evident seizures at 5-minute after starting study drug administration
Number of participants with sustained cessation of seizures | From 20 minutes to 60 minutes
  Number of participants with sustained cessation of clinically evident seizures from 20-minute to 60-minute after study drug administration with improved responsiveness (verbal communication, obeying commands, or purposeful reaction to painful stimuli) and no endotracheal intubation or use of any additional antiseizure medications or anticonvulsant sedatives.
Number of participants with recurrence of seizures | From 20 minutes to 4 hours
  Number of participants with recurrence of clinically evident seizures after initial control
Number of participants underwent endotracheal intubation | 60 minutes
  Number of participants underwent endotracheal intubation at 60 minutes after starting study drug administration
Number of participants with severe hypotension | 60 minutes
  Number of participants with severe hypotension at 60 minutes after starting study drug administration
Number of participants with severe hypertension | 60 minutes
  Number of participants with severe hypertension at 60 minutes after starting study drug administration
Number of participants with severe cardiac arrhythmia | 60 minutes
  Number of participants with severe cardiac arrhythmia at 60 minutes after starting study drug administration
Number of participants with emergence reactions | 4 hours
  Emergence reactions (hallucination, delirium, vivid dreams, blurred/double vision, hypersalivation) requiring benzodiazepines or other therapies within 4 hours after starting study drug administration
Number of participants admitted to Pediatric Intensive Care Unit | 24 hours
  Number of participants with admitted to Pediatric intensive Care Unit at 24 hours after starting study drug administration
Mortality | 24 hours
  All-cause mortality at 24 hours after starting study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics at Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
Unidentified individual participant data will be available to qualifying researchers upon a reasonable request